CLINICAL TRIAL: NCT06354062
Title: Talent Management Intervention Program for First Line Nurse Managers and Its Effect on Their Job Performance
Brief Title: Talent Management Intervention Program for First-Line Nurse Managers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Nagah Abd El-Fattah Mohamed Aly, Assistant professor of Nursing administration, Matrouh University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 0305896
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Intervention; Behavior; Knowledge, Attitudes, Practice
Keywords: Talent; Management,; Practice; Job Performance; Nurse Manager
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design
Who Masked: Participant
Masking Description: First Line Nurse Managers received talent Management intervention program
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of assistant head nurses (Other): First-line nurse managers received a talent management intervention program
  Interventions: Behavioral: Talent management intervention program
- Group of head nurses (Other): First-line nurse managers received a talent management intervention program
  Interventions: Behavioral: Talent management intervention program

INTERVENTIONS:
Behavioral: Talent management intervention program — Talent management intervention program

SUMMARY:
Nurse leaders will be required to manage the rapid change in the healthcare system. Talent management training plays a crucial role in preparing nursing leaders and improving their performance in health care systems.

DETAILED DESCRIPTION:
Nurse leaders will be required to manage the rapid change in the healthcare system. Talent management training plays a crucial role in preparing nursing leaders and improving their performance in health care systems. This study aimed to examine the effect of the talent management intervention program for first-line nurse managers on their job performance

ELIGIBILITY:
Inclusion Criteria:

* First-line nurse managers

  * willing to participate in the study
  * work in all inpatient care units of Alexandria University hospitals
  * Sign a consent

Exclusion Criteria:

* First-line nurse managers

  * work in outpatient units
  * Did not sign a consent
  * Absent from training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure nurse managers' knowledge | one month
  Knowledge of 125 nurse managers as assessed using a binary scale (0= No, 1= Yes). Change in nurse managers' knowledge level in one month
Questionnaire to measure talent management practice among first line nurse managers. | one month
  Talent management practice among first line nurse managers as assessed using five Likert scale (from 1= never and 5 = always).Change in nurse managers' practice in one month
Questionnaire to measure first-line nurse manager job performance | one month
  First-line nurse manager job performance as assessed using five Likert scale (1= Not once to 5= Always).Change in nurse managers' job performance in one month

CONTACTS AND LOCATIONS:
Overall Officials: Nagah Abd El-Fattah Mohamed Aly, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University, Egypt; Wael M. Lotfy, Ph.D, Study Director — Faculty of Nursing, Matrouh University, Egypt; Safaa M. El-Shanawany, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Maha Ghanem, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Faculty of Nursing, Matrouh University, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No